CLINICAL TRIAL: NCT06188442
Title: Superiority of On-demand Pre-exposure Prophylaxis Versus Post-exposure Prophylaxis on Using Doxycycline for Preventing Sexually Transmitted Infections in Men Who Have Sex With Men
Brief Title: Superiority of On-demand PrEP Versus PEP on Using Doxycycline for Preventing STI in MSM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz Ho Kwan, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23220262
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Sexually Transmitted Diseases, Bacterial; Syphilis; Gonorrhea; Chlamydia
Keywords: doxycycline; men who have sex with men; sexually transmitted infections
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial; Syphilis; Gonorrhea; Chlamydia Infections; Homosexuality; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: With a 3:1 intervention-to-control allocation ratio (198 and 66 participants would receive intervention and control, respectively), a total of 264 participants would be recruited.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DoxyODPrEP (Active Comparator): Participants in the DoxyODPrEP arm would be instructed to take two doxycycline hyclate 100mg capsules orally 2-24 hours before sex, and one 100mg capsule each 24 and 48 hours after loading dose. If they have sex within 48 hours after the loading dose, they would be asked to continue a daily 100mg until two days after the last sex.
  Interventions: Drug: DoxyODPrEP
- DoxyPEP (Active Comparator): Participants in the DoxyPEP arm would be instructed to take two doxycycline hyclate 100mg capsules orally within 24 hours and up to 72 hours after each sex.
  Interventions: Drug: DoxyPEP

INTERVENTIONS:
Drug: DoxyODPrEP — Participants in the DoxyODPrEP arm would be instructed to take two doxycycline hyclate 100mg capsules orally 2-24 hours before sex, and one 100mg capsule each 24 and 48 hours after loading dose. If they have sex within 48 hours after the loading dose, they would be asked to continue a daily 100mg until two days after the last sex
  Other Names: doxycycline on demand PrEP
  Arms: DoxyODPrEP
Drug: DoxyPEP — Participants in the DoxyPEP arm would be instructed to take two doxycycline hyclate 100mg capsules orally within 24 hours and up to 72 hours after each sex.
  Other Names: doxycycline PEP
  Arms: DoxyPEP

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of doxycycline taken for on-demand pre-exposure prophylaxis (DoxyODPrEP) and its post-exposure use (DoxyPEP) in preventing bacterial sexually transmitted infections (STI), including chlamydia, gonorrhoea, and syphilis among men who have sex with men (MSM). The main questions it aims to answer are:

1. Is DoxyODPrEP superior to DoxyPEP?
2. Are both regimens safe?
3. Does the MSM community accept the use of doxycycline to prevent bacterial STI?

Participants will be asked to take doxycycline according to the study arm they are randomly assigned to, and attend regular clinical follow-ups during the 2-year observation period. Researchers will compare the bacterial STI incidences between the two groups to see if DoxyODPrEP is superior to DoxyPEP.

DETAILED DESCRIPTION:
Participants would be randomly assigned to either DoxyODPrEP or DoxyPEP arm, and be instructed to take doxycycline with the respective dosing schedule. They would be followed up for 24 months for nucleic acid amplification test (NAAT) and antibody tests against bacterial STI, namely chlamydia, gonorrhoea, and syphilis. The subjects and investigators would not be blinded due to its open-label nature, as the two arms' dosing schedules are different. Participants in the DoxyODPrEP arm would be instructed to take two doxycycline hyclate 100mg capsules orally 2-24 hours before sex, and one 100mg capsule each 24 and 48 hours after loading dose. If they have sex within 48 hours after the loading dose, they would be asked to continue a daily 100mg until two days after the last sex. Participants in the DoxyPEP arm would be instructed to take two doxycycline hyclate 100mg capsules orally within 24 hours and up to 72 hours after each sex. At each clinic visit, urine, and pharyngeal and rectal swabs would be self-collected on-site by the participants following instructions. Pill count would be performed for each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* has had sex with another male in the past six months
* normally reside in Hong Kong
* can communicate in written and spoken Chinese or English
* willing and able to give written informed consent
* being willing and able to attend scheduled study clinic visits
* at risk of STI (had condomless sex with more than one man in the past 12 months, history of STI diagnosis in the past 12 months, inclination to have condomless sex, and other HIV-PrEP-eligible criteria)

Exclusion Criteria:

* Being allergic to tetracycline class medicines
* Currently taking medications that are contraindicated with doxycycline
* Using antibiotics for more than 14 days in the month preceding enrolment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to the first episode of gonorrhoea after the enrolment visit | Months 1 to 24
  Time to the first episode of gonorrhoea after the enrolment visit
Time to the first episode of chlamydia after the enrolment visit | Months 1 to 24
  Time to the first episode of chlamydia after the enrolment visit
Time to the first episode of syphilis after the enrolment visit | Months 1 to 24
  Time to the first episode of syphilis after the enrolment visit

SECONDARY OUTCOMES:
Safety profile | Months 1 to 24
  Percentage of participants experiencing adverse events and the associated grades
Acceptability of regimens | Months 1 to 24
  Percentage of participants accepted the regimen
Retention | Months 1 to 24
  Percentage of participants remained during the follow-up period
Time to the first episode of HIV after the enrolment visit | Months 1 to 24
  Time to the first episode of HIV after the enrolment visit

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ho Kwan, PhD, Principal Investigator — Jockey Club School of Public Health and Primary Care
Locations (1):
- Stanley Ho Centre for Emerging Infectious Diseases, Shatin, Hong Kong